CLINICAL TRIAL: NCT07069309
Title: A Phase 3 Protocol to Investigate the Safety, Tolerability, and Immunogenicity of BNT162b2 RNA-Based Variant-Adapted Vaccine Candidate(s) Against SARS-CoV-2 in Participants 12 Through 64 Years of Age Considered at Higher Risk of Severe COVID-19, and Participants ≥65 Years of Age
Brief Title: A Study to Learn About COVID-19 RNA-Based Variant-Adapted Vaccine Candidate(s) Against SARS-CoV-2 in Participants Ages 12 Through 64 Years Considered at Higher Risk of Severe COVID-19, and Participants Ages ≥65 Years
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: C4591076
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: COVID-19; SARS-COV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: 18 through 64 years of age (higher-risk individuals) (Experimental): Participants will receive BNT162b2 (2025/2026 recommended SARS-CoV-2 strain) 30 µg at Visit 1
  Interventions: Biological: BNT162b2 (2025/2026 recommended SARS-CoV-2 strain)
- Group 2: 65 years of age and older (Experimental): Participants will receive BNT162b2 (2025/2026 recommended SARS-CoV-2 strain) 30 µg at Visit 1
  Interventions: Biological: BNT162b2 (2025/2026 recommended SARS-CoV-2 strain)
- Group 3: 12 through 64 years of age (higher-risk individuals) (Experimental): Participants will receive BNT162b2 (2025/2026 recommended SARS-CoV-2 strain) 30 µg at Visit 1
  Interventions: Biological: BNT162b2 (2025/2026 recommended SARS-CoV-2 strain)
- Group 4: 65 years of age and older (Experimental): Participants will receive BNT162b2 (2025/2026 recommended SARS-CoV-2 strain) 30 µg at Visit 1
  Interventions: Biological: BNT162b2 (2025/2026 recommended SARS-CoV-2 strain)

INTERVENTIONS:
Biological: BNT162b2 (2025/2026 recommended SARS-CoV-2 strain) — BNT162b2 monovalent (2025/2026 recommended SARS-CoV-2 strain)

SUMMARY:
The purpose of this study is to learn about the safety, tolerability, and immunogenicity of an updated vaccine against COVID-19.

This study is seeking participants 12 through 64 years of age who are considered to be at higher risk for severe COVID-19 disease per study protocol and those 65 years of age and older. All participants in this study will receive 1 shot to their arm of a BNT162b2 (2025/2026 recommended SARS-CoV-2 strain) 30 µg RNA-based vaccine which targets a circulating variant of SARS-CoV-2 and is selected for the 2025-2026 COVID-19 respiratory virus season. This study is about 6 months for each participant. Participants will either be enrolled in Cohort 1 (Groups 1 and 2) or Cohort 2 (Groups 3 and 4). Participants enrolled in Cohort 1 will have at least 4 visits and participants enrolled in Cohort 2 will have at least 3 visits.

ELIGIBILITY:
Inclusion criteria:

* Cohort 1: Participants 18 years of age or older.
* Cohort 2: Participants 12 years of age or older.
* Participants 12 through 64 years of age with at least 1 underlying medical condition that increases their risk of severe COVID-19.

Exclusion Criteria:

* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s).
* History of myocarditis or pericarditis.
* Cohort 2: Receipt of a COVID-19 vaccine or a confirmed case of COVID-19 (confirmed by signs/symptoms and/or a positive test result based on local testing) less than 5 months (150 days) prior to study enrollment.

Refer to the study contact for further eligibility details.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 760 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2026-05-05 (Estimated); Study Completion 2026-05-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants reporting local reactions | For up to 7 days after vaccination
Percentage of participants reporting systemic events | For up to 7 days after vaccination
Percentage of participants reporting adverse events | Through 1 month after vaccination
Percentage of participants reporting serious adverse events | Through 6 months after vaccination
Cohort 1: Geometric Mean Titers (GMTs) | At 2 weeks after vaccination
Cohort 1: Geometric Mean Fold Rises (GMFRs) | From before vaccination to 2 weeks after vaccination
Cohort 1: Percentages of participants with seroresponse | 2 weeks after vaccination
Cohort 2: Geometric Mean Fold Rises (GMFRs) | From before vaccination to 1 month after vaccination

SECONDARY OUTCOMES:
Cohort 1: Geometric Mean Titers (GMTs) | At 1 month after vaccination
Cohort 1: Geometric Mean Fold Rises (GMFRs) | From before vaccination to 1 month after vaccination
Cohort 1: Percentages of participants with seroresponse | 1 month after vaccination
Cohort 2: Geometric Mean Titers (GMTs) | From before vaccination to 1 month after vaccination
Cohort 2: Percentages of participants with seroresponse | 1 month after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- United States (19):
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Clinical Research Consulting, Milford, Connecticut
  - GW Vaccine Research Unit, Washington D.C., District of Columbia
  - The GW Medical Faculty Associates, Washington D.C., District of Columbia
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Palm Springs Community Health Center, Miami Lakes, Florida
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Kentucky Pediatric/ Adult Research, Bardstown, Kentucky
  - Bio-Kinetic Clinical Applications, LLC dba QPS-MO, Springfield, Missouri
  - Bio-Kinetic Clinical Applications, LLC dba QPS-MO-Screening and Recruitment Center, Springfield, Missouri
  - Rochester Clinical Research, LLC, Rochester, New York
  - Accellacare - Wilmington, Wilmington, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Senders Pediatrics, South Euclid, Ohio
  - DM Clinical Research - Philadelphia, Philadelphia, Pennsylvania
  - DM Clinical Research- Cyfair, Houston, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591076